CLINICAL TRIAL: NCT01323595
Title: The Use of Celecoxib (Celebrex (c)) in Post-operative Pain Control After Microdissection Testicular Sperm Extraction
Brief Title: Effectiveness of Celecoxib After Surgical Sperm Retrieval
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Interim analysis demonstrated significant benefit in intervention arm
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1010011319
Record Dates: First submitted 2011-03-24; First posted 2011-03-25 (Estimated); Results first posted 2014-07-11 (Estimated); Last update posted 2018-10-02 (Actual); Status verified 2018-09

CONDITIONS: Pain
Keywords: Pain control; testicular sperm extraction; sperm
MeSH Terms: conditions — Pain; Agnosia | interventions — Celecoxib; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Celecoxib (Experimental): Celecoxib will be given for 6 days after surgery
  Interventions: Drug: Celecoxib
- Sugar pill (Placebo Comparator): Sugar pill for 6 days after surgery.
  Interventions: Drug: Sugar Pill

INTERVENTIONS:
Drug: Celecoxib — Celecoxib 200mg PO BID x 6 days
  Other Names: Celebrex
  Arms: Celecoxib
Drug: Sugar Pill — Sugar pill PO BID x 6 days
  Other Names: Placebo
  Arms: Sugar pill

SUMMARY:
While narcotic medication are commonly used for pain control near the time of surgery, there are significant side effects including constipation, nausea, risk of overdose leading to decreased breathing, and risk of addiction to narcotics. Our goal is to explore alternatives to narcotics for perioperative pain for patients undergoing sperm retrieval surgery. We have designed a prospective randomized clinical trial to evaluate how effective the anti-inflammatory medicine celecoxib(Celebrex©) is for pain control near the time of surgery. Celecoxib is known as a COX-2 inhibitor, a drug that belongs to the non-steroidal anti-inflammatory drug (NSAID) class. It is used to reduce swelling and to treat pain.

Patients will be divided into two groups: the first group receives a celecoxib pill and the second group receives a sugar pill(placebo). Patients and doctors will be unaware of exactly which pills are given. The patient will complete questionnaires for pain level. By comparing the pain levels we can better understand whether celecoxib (Celebrex©) significantly decreases perioperative pain.

DETAILED DESCRIPTION:
All consecutive patients scheduled to undergo elective, outpatient microsurgical testicular sperm extraction (TESE) beginning in 9/2011 will be invited for participation. Microdissection TESE will be performed unilaterally or bilaterally, through a midline scrotal incision, under general anesthesia.

Participants will be prospectively randomized in a 1:1 ratio to receive 200 mg of celecoxib or placebo b.i.d. in a double-blind fashion, initiated the night prior to surgery, and continued for six days thereafter. The randomization sequence will be generated and implemented by the institutional investigational pharmacy. Placebo medication, identical to the study medication, will also be provided by the institutional pharmacy.

Following surgery, all participants will be asked to complete a take-home post-operative questionnaire recording their maximum pain level on an 11-point visual analog scale (0-10), at specific time intervals over the course of the day, ranging from every six hours on post-operative day (POD) #1 to every 8 hours on POD #2, every 12 hours on POD #3, and every 24 hours on POD #4 to POD #7. Patients will also record the number of 5/500 mg tablets of acetaminophen/hydrocodone used for supplemental pain control from POD #1 to POD #7. Thirdly, patients will record whether or not their pain was adequately controlled at each of the above-mentioned time intervals.

ELIGIBILITY:
Inclusion Criteria:

1. >/= 18 years old
2. Male
3. Scheduled to undergo microdissection testicular sperm extraction

Exclusion Criteria:

1. History of allergies to celecoxib (Celecoxib)
2. Renal failure
3. History of ulcer disease
4. Any history of myocardial infarction
5. Any history of stroke
6. History of bleeding diathesis
7. Use of aspirin

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2011-01; Primary Completion 2012-12 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter N Schlegel, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Department of Urology, Weill Cornell Medical College,, New York, New York, United States

REFERENCES:
- See also: Study Abstract — http://www.ncbi.nlm.nih.gov/pubmed/23628190

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients undergoing testicular sperm extraction surgery
Pre-assignment Details: No exclusions except allergy to treatment agent (celecoxib)
Groups:
- Celecoxib: Celecoxib will be given for 5 days after surgery
  Celecoxib : Celecoxib 200mg PO BID x 6 days
- Sugar Pill: Sugar pill for 5 days after surgery.
  Sugar Pill : Sugar pill PO BID x 6 days
Period: Overall Study
Arm/Group | Celecoxib | Sugar Pill
Started | 39 | 39
Completed | 16 (Remaining subjects did not return questionnaire) | 18 (Remaining subjects did not return questionaire)
Not Completed | 23 | 21

BASELINE CHARACTERISTICS:
Groups:
- Celecoxib: Celecoxib will be given for 6 days after surgery
  Celecoxib : Celecoxib 200mg PO BID x 6 days
- Sugar Pill: Sugar pill for 6 days after surgery.
  Sugar Pill : Sugar pill PO BID x 6 days
- Total: Total of all reporting groups
Arm/Group | Celecoxib | Sugar Pill | Total
Number analyzed (Participants) | 39 | 39 | 78
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 39 | 39 | 78
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 39 (5) | 35 (5) | 37 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 39 | 39 | 78
Region of Enrollment [Number; unit: participants]
  United States | 39 | 39 | 78

OUTCOME MEASURES:

1. Primary Outcome: Level of Pain
Description: Patients will rate their pain for 7 days after surgery using an 11-point visual analog scale, ranging from 0 to 10, in which 0= no pain, 10=worst pain ever. Patients are asked to rate their pain up to four times a day during the post-operative period. Pain scores from each post-operative day each day will be averaged and reported as the pain score for that day.
Time Frame: 1 week after surgery
Measure: Mean (Standard Deviation); unit: Analog pain scale
Groups:
- Placebo Treatment: Patients received placebo medication
- Celecoxib: Patients received celecoxib
Arm/Group | Placebo Treatment | Celecoxib
Number analyzed (Participants) | 18 | 16
Analog pain scale | 6 (2) | 4 (2)

2. Secondary Outcome: Number of Participants With Bleeding Complications
Description: We will record whether there are any bleeding complications associated with treatment after surgery.
Time Frame: 7 days after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Celecoxib | Sugar Pill
Number analyzed (Participants) | 16 | 18
Participants | 0 | 0

ADVERSE EVENTS:
Arm/Group | Placebo Treatment | Celecoxib
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/16
Other Adverse Events (participants affected / at risk) | 0/18 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No